CLINICAL TRIAL: NCT01397617
Title: Evaluation of NobelBiocare SFB and CFB Implants
Brief Title: Randomized, Open Investigation Evaluating the Efficacy of Nobel Biocare SFB and CFB Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-117
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Partial Edentulism; Complete Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NobelActive Internal (Experimental): NobelActive Internal implant
  Interventions: Device: NobelActive Internal implant
- NobelActive External (Experimental): NobelActive External implant
  Interventions: Device: NobelActive External implant
- NobelReplace Tapered Groovy (Active Comparator): NobelReplace Tapered Groovy implant
  Interventions: Device: NobelReplace Tapered Groovy implant

INTERVENTIONS:
Device: NobelActive Internal implant — Dental implant
  Arms: NobelActive Internal
Device: NobelActive External implant — Dental implant
  Arms: NobelActive External
Device: NobelReplace Tapered Groovy implant — Dental implant
  Arms: NobelReplace Tapered Groovy

SUMMARY:
The purpose of this study is to determine the survival rate, marginal bone resorption, soft tissue health and maintenance of the NobelActive Internal and External implants and to make comparisons with the NobelReplace Tapered Groovy implant placed in healed sites.

DETAILED DESCRIPTION:
The purpose of this study is to determine safety and efficacy parameters for the NobelActive Internal and External implants and to make comparisons with the NobelReplace Tapered Groovy implant placed in healed sites.

Safety: AEs

Efficacy:

* survival rates,
* marginal bone resorption with marginal bone levels measurement,
* soft tissue health and maintenance via gingival index measurement, plaque index, papilla index .

ELIGIBILITY:
Inclusion Criteria:

* The subject should be in need of an implant supported fixed restoration
* The subjects should have sufficient bone volume and density i.e. an osseous architecture in the planned implant placement region sufficient to receive implants with a diameter of 3.5 mm and a length of at least 10 mm.
* The subject as well as the implant sites should fulfill criteria for immediate functional tem-porization within 24 h.
* The implant sites should be healed and free from infection.

Exclusion Criteria:

* Alcohol or drug abuse as noted in patient records or in patient history.
* Health conditions, which do not permit the surgical procedure.
* Reason to believe that the treatment might have a negative effect on the subject's total situation (psychiatric problems), as noted in patient records or in patient history.
* The subject is not able to give her/his informed consent to participate.
* The need of bone augmentation before implant installation to obtain a prosthetically correct implantation transversally. However, a minor augmentation procedure to cover exposed threads or interproximal / buccal grafting due to deficient sites is not an exclusion criteria.
* Any disorders in the planned implant area such as previous tumors, chronic bone disease, or previous irradiation.
* Uncontrolled diabetics will be excluded.
* Severe bruxism or other destructive habits.
* Immediate insertion (e.g. placement of the implant immediately after extraction) consti-tutes an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2006-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnhart C, Kielbassa AM, Martinez-de Fuentes R, Goldstein M, Jackowski J, Lorenzoni M, Maiorana C, Mericske-Stern R, Pozzi A, Rompen E, Sanz M, Strub JR. Comparison of variable-thread tapered implant designs to a standard tapered implant design after immediate loading. A 3-year multicentre randomised controlled trial. Eur J Oral Implantol. 2012 Summer;5(2):123-36. PMID 22866289

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NobelActive Internal | NobelActive External | NobelReplace Tapered Groovy
Started | 64 | 53 | 60
Completed | 33 | 30 | 31
Not Completed | 31 | 23 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NobelActive Internal | NobelActive External | NobelReplace Tapered Groovy | Total
Number analyzed (Participants) | 64 | 53 | 60 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.1) | 49.9 (13.6) | 46.9 (14.6) | 48.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 21 | 34 | 92
  Male | 27 | 32 | 26 | 85

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Was the Change in Marginal Bone Levels (in mm) From the Time of Implant Insertion to Follow-up Visits (3,6,12,24,36 and 60 Months).
Description: Marginal bone remodeling is calculated for each side of the implant (mesial and distal) separately, as the difference between bone levels at two time points. The average of mesial and distal remodeling is then calculated for each implant site (paired for each side between two different points). Negative numbers indicate bone loss. Implant insertion was defined as a baseline.
  Missing data was not imputed and not included in evaluation.
Time Frame: baseline, 3 months, 6 months, 12 months, 24 months, 36 months and 60 months
Population: Intent to treat analysis (all participants who received at least one implant were analyzed). Missing data was not imputed and not included in evaluation.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | NobelActive External | NobelActive Internal | NobelReplace Tapered Groovy
Number analyzed (Participants) | 53 | 64 | 60
mm
  implant insertion to 60 months | -0.31 (1.50) | -0.98 (1.60) | -1.13 (1.67)
  implant insertion to 36 months | -0.16 (1.06) | -0.89 (1.65) | -0.85 (1.32)
  implant insertion to 24 months | -0.35 (0.83) | -0.68 (1.35) | -0.96 (1.25)
  implant insertion to 12 months | -0.64 (0.97) | -0.95 (1.37) | -0.63 (1.17)
  implant insertion to 6 months | -0.92 (0.96) | -1.03 (1.36) | -0.75 (1.13)
  implant insertion to 3 months | -0.95 (1.03) | -0.96 (1.15) | -0.86 (0.99)

2. Secondary Outcome: Implant Survival Rate From the Time of Implant Insertion to Follow-up Visits (3,6,12,24,36 and 60 Months).
Description: An implant was reported to be a surviving implant when it remained in the jaw and was functionally loaded even if not all the individual success criteria were fulfilled (i) an implant that causes no allergic, toxic or gross infectious reactions either locally or systemically, ii) offered anchorage to a functional prosthesis, iii) showed no signs of fracture or bending, iv) showed no signs of peri-implant radiolucency on an intraoral radiograph using a paralleling technique strictly perpendicular to the implant-bone interface, and v) showed no mobility when individually tested by either tapping or rocking with a hand instrument).
Time Frame: baseline, 3 months, 6 months, 12 months, 24 months, 36 months and 60 months
Population: Intention to treat analysis.
Measure: Number; unit: percentage of surviving implants
Units Other Than Participants: implants
Arm/Group | NobelActive Internal | NobelActive External | NobelReplace Tapered Groovy
Number analyzed (Participants) | 64 | 53 | 60
Number analyzed (implants) | 117 | 82 | 126
percentage of surviving implants
  60 months | 94.6 | 96.3 | 96.6
  36 months | 95.7 | 96.3 | 96.6
  24 months | 95.7 | 96.3 | 97.6
  12 months | 96.6 | 96.3 | 97.6
  6 months | 98.3 | 96.3 | 97.6
  3 months | 98.3 | 97.6 | 98.4

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the duration of the study with the 5-year follow up.
Description: From implant insertion to 5 years follow-up 31 patient was lost to follow-up in NobelActive External group, 31 patient was lost to follow-up in NobelActive Internal group and 29 patient was lost to follow-up in NobelReplace group.
Arm/Group | NobelActive External | NobelActive Internal | NobelReplace Tapered Groovy
Serious Adverse Events (participants affected / at risk) | 2/30 | 1/33 | 3/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NobelActive External (N=30) | NobelActive Internal (N=33) | NobelReplace Tapered Groovy (N=31)
stroke (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute leukemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
cardiac valve surgery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypesthesia (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
squamous cell cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No